CLINICAL TRIAL: NCT03538925
Title: Word by Word: Building Sentences With Preschoolers Who Use AAC
Brief Title: Building Sentences With Preschoolers Who Use AAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Central Florida (Other)
Collaborators: University of New Mexico (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1061417; R01DC016321 (NIH)
Record Dates: First submitted 2018-05-16; First posted 2018-05-29 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Down Syndrome; Speech and Language Disorder; Speech Disorders in Children; Speech Intelligibility; Speech Sound Disorder
MeSH Terms: conditions — Down Syndrome; Speech; Language Disorders; Speech Intelligibility; Speech Sound Disorder | interventions — Standard of Care; Commerce

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): AAC Generative Language Intervention
  Interventions: Behavioral: AAC Generative Language Intervention; Behavioral: Standard of Care / Business as Usual
- Business as Usual (Active Comparator): Standard of Care / Business as Usual
  Interventions: Behavioral: Standard of Care / Business as Usual

INTERVENTIONS:
Behavioral: AAC Generative Language Intervention — Parent/Caregiver AAC App Operational Training + Direct AAC Input-Output Language Intervention
  Arms: Treatment Group
Behavioral: Standard of Care / Business as Usual — Parent/Caregiver AAC App Operational Training

SUMMARY:
The focus of this investigation is to compare the effectiveness of the AAC Generative Language Intervention approach to an AAC Standard of Care condition on preschool sentence productions. All children will use existing AAC iPad applications.

DETAILED DESCRIPTION:
The central hypothesis is that preschoolers receiving AAC Generative Language Intervention will create longer, more grammatically complete sentences compared with the Standard of Care condition. Specific Aim 1 compares these interventions for preschoolers with severe speech impairments and typical receptive language, and Specific Aim 2 does the same for children with Down syndrome. Specific Aim 3 tests for possible moderation of the intervention effect by age, dynamic assessment scores, sentence type, receptive language abilities, prior AAC use, sex, mental age, and disability. Aims 1 and 2 will be accomplished using randomized controlled trials.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Identification of Significant Speech Impairment
* Must Speak English as a Primary Language
* Must Be Able to Express At Least 25 Words (using any communication mode)
* Must Be Able to Accurately Select Picture Symbols on iPad Communication App with at Least 50% Accuracy
* Vision and Hearing within Functional Limits or Corrected to be within Functional Limits for Study Activities

Exclusion Criteria:

* Clinical Diagnosis of Autism or Social Communication Disorder
* Primary Language Spoken is a Language Other than English

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2018-05-11 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Aided AAC Utterance Length | 6 Months
  Aided AAC sentence length measured in morphemes

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - FAAST Center at the University of Central Florida, Orlando, Florida
  - University of New Mexico Department of Speech and Hearing Sciences, Albuquerque, New Mexico

IPD SHARING:
Plan to Share IPD: No